CLINICAL TRIAL: NCT05887583
Title: Supporting Physical Literacy at School and Home (SPLASH) Study
Brief Title: Supporting Physical Literacy at School and Home
Acronym: SPLASH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: George Washington University (Other)
Responsible Party: Principal Investigator, Erin Hennessy, Assistant Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003794
Record Dates: First submitted 2023-05-10; First posted 2023-06-02 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-01

CONDITIONS: Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Schools will be randomized to receive either the intervention or control group condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The Rising New York Road Runners program: A School-based physical education curriculum with family engagement component.
  Interventions: Behavioral: The Rising New York Road Runners program
- Control (No Intervention): Standard school operating procedures

INTERVENTIONS:
Behavioral: The Rising New York Road Runners program — The Rising New York Road Runners program provides lesson plans covering fundamental movement skills that are intended to build competence, confidence, and motivation to be physically activity. Family engagement materials (emails, text messages, videos, social media) complement school materials to communicate what children are learning at school related to physical activity and what activities families can do at home together to reinforce these concepts.
  Other Names: Rising New York Road Runners
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to test if a multilevel (school, home) physical activity intervention for school-aged (3rd-5th grade) children can increase physical activity levels. The main question[s] it aims to answer are:

* The impact of the multilevel program on children's physical literacy and physical activity over one school year. Hypothesis:
* Whether the program effects are different by children's gender or weight status
* Whether changes in children's ability, confidence and motivation for physical activity are related to changes in physical activity levels.

Schools will be randomly assigned to receive the multilevel intervention or a control group.

Participants in the intervention group will receive a new school curriculum during regular physical education classes and information for families on what school activities can be done at home.

Researchers will compare outcomes according to intervention and control group assignments.

DETAILED DESCRIPTION:
Low levels of physical activity (PA) among youth remain a significant public health problem, with most U.S. children falling short on the recommended 60 minutes of daily moderate-to-vigorous physical activity (MVPA). Research shows that this gap disproportionately affects population subgroups, particularly children who are female, overweight/obese, or from low socioeconomic areas. Interventions are needed that can equitably increase children's PA. To address this gap, there has been a focus in the U.S. and abroad on increasing children's physical literacy (PL), which can be defined as the ability, confidence, and motivation to be physically active for life. While PL-focused interventions hold promise in concept, there is little empirical evidence of effectiveness and differential effects by subgroups are not understood. Thus, the overall objective is to increase children's PA through a multilevel, comprehensive PL-focused program that will reach children both at school and at home. The overarching hypothesis is that the PL-focused program will have positive effects on elementary schoolchildren's PL and, in turn, PA.

Aims include testing the multilevel Rising New York Road Runners (RNYRR) program using a 2-arm, group randomized controlled trial (RCT) with n=400 3rd-5th grade students from low-income schools receiving either the multilevel RNYRR program (n=4) or delayed-intervention control (n=4).

Aim 3: To evaluate the impact of the RNYRR program on children's physical literacy (PL) and physical activity (PA) (total daily volume and moderate-to-vigorous PA (MVPA)) over one school year. Hypothesis: Children who attend schools with the RNYRR programming will increase PL and PA (total daily volume and MVPA) relative to children in control schools.

Aim 3a: To examine whether RNYRR program effects on children's PL and PA differ by sex or weight status.

Aim 3b: To test whether changes in PL and PL subdomains (e.g. ability, confidence, motivation) mediate changes in daily total PA volume or MVPA.

ELIGIBILITY:
Inclusion Criteria:

* Child attends school participating in the intervention
* In the 3rd, 4th or 5th grade
* Participates in the school's physical education class

Exclusion Criteria:

* Not in the 3rd, 4th or 5th grade
* Does not participate in the school's physical education class

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Baseline physical activity level | +/- 4 weeks prior to study intervention
  Children will wear an Actigraph accelerometer for 7 days on their right hip at study baseline (prior to intervention). The accelerometer measures vertical acceleration across three planes and computes a total volume of movement over a specified amount of time set by the researcher. This information will also be used to computer time spent in intensity-specific physical activity using established cutpoints.
End-point physical activity level | +/- 4 weeks prior to study completion
  Children will wear an Actigraph accelerometer for 7 days on their right hip at study baseline (prior to intervention). The accelerometer measures vertical acceleration across three planes and computes a total volume of movement over a specified amount of time set by the researcher. This information will also be used to computer time spent in intensity-specific physical activity using established cutpoints.

SECONDARY OUTCOMES:
Baseline fundamental movement skill in running, locomotion, object control and Balance | +/- 4 weeks prior to study intervention
  Trained staff will administer the Physical Literacy Assessment for Youth tool to assess children's performance across 18 different tasks that assess competence in fundamental movement skill domain areas: Running, locomotion, object control and balance.
End-point fundamental movement skill in running, locomotion, object control and Balance | +/- 4 weeks prior to study completion
  Trained staff will administer the Physical Literacy Assessment for Youth tool to assess children's performance across 18 different tasks that assess competence in fundamental movement skill domain areas: Running, locomotion, object control and balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
No.